CLINICAL TRIAL: NCT00428714
Title: Phase 2 Trial Oral Enzastaurin in Prostate Cancer Patients Who Have Rising PSA (1) During Hormonal Manipulation and (2) After First-Line Cytotoxic Chemotherapy
Brief Title: Phase 2 Trial of Enzastaurin in Prostate Cancer in Participants Who Have Had Hormonal and Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10737; H6Q-MC-S024 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enzastaurin-Cohort 1 (Experimental): Chemo-naive participants who had androgen-independent prostate cancer with rising prostate-specific antigen (PSA) levels but no clinical or radiographic evidence of metastatic disease. Participants were given 1125 mg loading dose of enzastaurin on Day 1 of Cycle 1 (28-day cycle) only, and thereafter 500 mg enzastaurin once daily.
  Interventions: Drug: enzastaurin
- Enzastaurin-Cohort 2 (Experimental): Participants with progressed, metastatic prostate cancer who had received prior treatment with a docetaxel-containing agent. Participants were given 1125 mg loading dose of enzastaurin on Day 1 of Cycle 1 (28-day cycle) only, and thereafter 500 mg enzastaurin once daily.
  Interventions: Drug: enzastaurin

INTERVENTIONS:
Drug: enzastaurin — Administered orally
  Other Names: LY317615

SUMMARY:
The purpose is to see how quickly two different types of prostate cancer participants respond when taking enzastaurin.

Cohort 1 - asymptomatic participants with androgen-independent prostate-specific antigen (PSA)-progressive disease without clinical or radiographic evidence of metastatic disease.

Cohort 2 - participants with androgen-independent metastatic prostate cancer (documented bone or soft tissue metastases) with rising PSA, clinical, radiographic disease progression following one prior docetaxel-based regimen

ELIGIBILITY:
Inclusion Criteria:

* You are expected to be alive in the 12 weeks.
* You are at least 18 years old.
* You live close enough to the doctor's office to attend all of your required visits.
* You have not been treated with chemotherapy for your prostate cancer (cohort 1).
* Must have evidence of androgen-independent PSA-progressive disease without a history of or current (as judged by the investigator) clinical or radiographic evidence of metastatic disease with castrate levels of testosterone (<50 ng/dL) maintained by luteinizing hormone-releasing hormone (LHRH) agonist or bilateral orchiectomy following standard anti-androgen withdrawal. NOTE: PSA progression is defined as have rising PSA values of <=5 ng/mL (at least 3 measurements 1 week apart) with castrate levels of testosterone <50 ng/dL following appropriate antiandrogen withdrawal, without evidence of metastases. (cohort 1)
* No prior systemic chemotherapy for prostate cancer. No prior chemotherapy for any other indication within 2 years of study entry. NOTE: Participants previously treated with chemotherapy in the adjuvant/neoadjuvant setting were not be eligible. (cohort 1)
* You have had one prior docetaxel-based chemotherapy regimen (cohort 2).
* You have evidence of metastatic prostate cancer with bone or soft tissue disease (cohort 2).
* Must have evidence of docetaxel-resistant, androgen-independent metastatic prostate cancer with bone or soft tissue disease (PSA only participants are not eligible) defined as either: clinical, PSA or radiographic disease progression while receiving docetaxel-based therapy or PSA and/or radiographic progression at any time after completion of a docetaxel-containing regimen with PSA progression defined as a 25% increase in PSA from the post docetaxel value or interval progression in known metastatic sites of disease or development of new sites of disease on bone scan or computed tomography (CT) imaging. Note: Participants who discontinued a docetaxel-containing regimen due to toxicity or any other reasons not related to disease progression while on treatment, and were not able to complete at least 2 cycles, were not be eligible. (cohort 2)
* Your organs must be functioning properly.

Exclusion Criteria:

* You are unable to swallow pills.
* You have another illness besides your prostate cancer.
* You have taken another experimental drug within the last 30 days.
* You have a serious heart condition.
* You are receiving another anti-cancer therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stanford, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buffalo, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin

REFERENCES:
- [Derived] Dreicer R, Garcia J, Hussain M, Rini B, Vogelzang N, Srinivas S, Somer B, Zhao YD, Kania M, Raghavan D. Oral enzastaurin in prostate cancer: a two-cohort phase II trial in patients with PSA progression in the non-metastatic castrate state and following docetaxel-based chemotherapy for castrate metastatic disease. Invest New Drugs. 2011 Dec;29(6):1441-8. doi: 10.1007/s10637-010-9428-0. Epub 2010 Apr 6. PMID 20369375
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Table presents reason for treatment discontinuation.
Groups:
- Enzastaurin-Cohort 1: Chemo-naive participants who had androgen-independent prostate cancer with rising PSA levels but no clinical or radiographic evidence of metastatic disease. Participants were given 1125 mg loading dose of enzastaurin on Day 1 of Cycle 1 (28-day cycle) only, and thereafter 500 mg enzastaurin once daily.
Period: Overall Study
Arm/Group | Enzastaurin-Cohort 1 | Enzastaurin-Cohort 2
Started | 31 | 42
Received at Least 1 Dose of Study Drug | 31 | 42
Completed | 0 | 0
Not Completed | 31 | 42
Not completed — Progressive Disease | 28 | 36
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Death due to Progressive Disease (PD) | 1 | 0
Not completed — Death due to other then PD | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Enzastaurin-Cohort 1 | Enzastaurin-Cohort 2 | Total
Number analyzed (Participants) | 31 | 42 | 73
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 72.2 (10.0) | 69.9 (7.77) | 70.88 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 31 | 42 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27 | 39 | 66
  African | 3 | 0 | 3
  Hispanic | 1 | 1 | 2
  East Asian | 0 | 1 | 1
  West Asian | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 42 | 73
Eastern Cooperative Oncology Group Scale Performance Status (ECOG) [Count of Participants; unit: Participants] — Classifies participants according to their functional impairment. Scores range from 0 (Fully Active), 1 (ambulatory with restricted strenuous activity), 2 (ambulatory, no work activities), to 5 (Death).
  Participants
    0 | 22 | 14 | 36
    1 | 9 | 26 | 35
    2 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1 - Number of Participants With a Complete Response (CR) or Partial Response (PR) (Objective Response Rate)
Description: Objective responders were defined as participants (pts) in Cohort 1 who met prostate-specific antigen (PSA) response criteria. PSA Complete response (CR) was defined as a decrease in PSA to an undetectable level (<0.2 ng/mL) confirmed by a second value obtained at least 4 weeks apart and without clinical or radiographic evidence of disease. PSA Partial Response (PR) was defined as a decrease in PSA of >=50% at any time during the study. The decline of >=50% in PSA must be from a baseline value of >5 ng/mL and must be confirmed by a second value obtained at least 4 weeks apart and without clinical or radiographic evidence of disease.
Time Frame: Baseline to Measured Progressive Disease, Death, Unacceptable Toxicities, or Study Closure Whichever Occurred First (up to 56 weeks)
Population: Participants in Cohort 1 with a valid baseline and at least one post-baseline PSA assessment.
Measure: Number; unit: Participants
Arm/Group | Enzastaurin-Cohort 1
Number analyzed (Participants) | 27
Participants | 1

2. Primary Outcome: Cohort 2 - Progression-free Survival (PFS)-Overall
Description: PFS was defined as the time from date of enrollment to first occurrence of (1) tumor progression (defined per Response Evaluation Criteria In Solid Tumors [RECIST]) for soft tissue lesions, and/or appearance of >=2 new lesions on bone scan (confirmed >=6 weeks later); (2) skeletal event (pathological bone fracture and/or need for palliative radiotherapy); (3) symptomatic progression (worsening of Eastern Cooperative Oncology Group (ECOG) performance status (PS) and/or weight loss >10% from baseline and/or increase in analgesic consumption and pain); or (4) Death due to any cause. PFS was censored at date of last objective progression-free observation for participants who were still alive and had not progressed. Participants who took any subsequent systemic anticancer therapy prior to progression or death were censored at date of last objective progression-free disease assessment prior to the date of the subsequent systemic anticancer therapy.
Time Frame: baseline to first occurrence of tumor progression, skeletal event, symptomatic progression, or death (up to 31.3 weeks)
Population: Participants in Cohort 2 who received at least 1 dose of enzastaurin. Two participants were censored.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Enzastaurin-Cohort 2
Number analyzed (Participants) | 42
Weeks | 11.0 [7.57 to 11.7]

3. Secondary Outcome: Cohort 1 - Number of Participants With a 3-month PSA Level Decline of Greater Than or Equal to 30%
Description: Number of participants exhibiting a PSA level decline from baseline of greater than or equal to 30% within the first 3 months of study.
Time Frame: baseline to 3 months
Population: Participants Cohort 1 with a valid baseline and at least one post-baseline PSA assessment.
Measure: Number; unit: participants
Arm/Group | Enzastaurin-Cohort 1
Number analyzed (Participants) | 27
participants | 1

4. Secondary Outcome: Cohort 1 - PSA Velocity
Description: PSA velocity is defined as the rate of change in the PSA level during the first 2 and 3 months of the study.
Time Frame: baseline, 2 months and 3 months
Population: Participants in Cohort 1 with a valid baseline and at least one post-baseline PSA measurement within the first 2 and 3 months of treatment, respectively.
Measure: Mean (Full Range); unit: nanograms per milliliter per year
Groups:
- LY317615- Cohort 1: Chemo-naive participants who had androgen-independent prostate cancer with rising PSA levels but no clinical or radiographic evidence of metastatic disease. Participants were given 1125 mg loading dose of enzastaurin on Day 1 of Cycle 1 (28-day cycle) only, and thereafter 500 mg enzastaurin once daily.
Arm/Group | LY317615- Cohort 1
Number analyzed (Participants) | 27
nanograms per milliliter per year
  PSA Velocity at 2 months | 0.10003 [-1.6080 to 0.59390]
  PSA Velocity at 3 months | 0.06289 [-2.5093 to 0.51271]

5. Secondary Outcome: Cohort 1 - Progression-free Survival (PFS)-Overall
Description: Progression free survival (PFS) is defined as the time from the date of enrollment to the first occurrence of PSA progression or objective progression defined as development of radiographic evidence of metastatic disease irrespective of PSA value or death due to any cause. PSA progression is defined as (a) for participants in whom a 50% decline in PSA has not been achieved, this is defined as 25% increase over baseline or nadir whichever is lower and an increase in the absolute value of PSA level by 5 ng/mL that is confirmed by another value of PSA confirmed at least 4 weeks apart; (b) for participants in whom a 50% decline in PSA has been achieved, this is defined as 50% increase over the nadir and an increase in the absolute value of PSA level by 5 ng/mL that is confirmed by another PSA level at least 4 weeks apart.
Time Frame: baseline to date of disease progression, death, unacceptable toxicities, or study closure whichever occurred first (up to 56 weeks)
Population: Participants in Cohort 1 with a valid baseline and at least one post-baseline PSA assessment. Two participants were censored.
Measure: Median (Full Range); unit: weeks
Arm/Group | Enzastaurin-Cohort 1
Number analyzed (Participants) | 27
weeks | 12 [4 to 56]

6. Secondary Outcome: Cohort 1 - Duration of Response
Description: Duration of response was the date of first objective assessment of CR or PR to the date of first progression or death due to any cause. Progression of disease defined as:1) PSA progression: (a) in whom a 50% decline in PSA has not been achieved, defined as 25% increase over baseline or nadir whichever is lower and an increase in the absolute value of PSA level by 5 ng/mL and confirmed by another PSA at least 4 weeks apart, (b) in whom a 50% decline in PSA has been achieved, defined as 50% increase over the nadir and an increase in the absolute value of PSA level by 5 ng/mL and confirmed by another PSA level at least 4 weeks apart. 2) Objective Progression defined as radiographic evidence of metastatic disease irrespective of PSA value or 3) death due to any cause. Duration of response was censored on the date of discontinuation or last assessment for those participants who were alive without progression.
Time Frame: time of response to progressive disease, death, unacceptable toxicities, or study closure whichever occurred first (up to 56 weeks)
Population: Participants in Cohort 1 with a CR or PR who had a valid baseline and at least one post-baseline PSA assessment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Enzastaurin-Cohort 1
Number analyzed (Participants) | 1
weeks | 27.9 [NA to NA] — 95% confidence interval was not estimable as only one participant had response.

7. Secondary Outcome: Cohort 2 - 3-month PSA Level Decline of Greater Than or Equal to 30%
Description: as for outcome 3
Time Frame: baseline to 3 months
Population: Participants in Cohort 2 with a valid baseline and at least one post-baseline PSA measurement within the first 3 months of treatment.
Measure: Number; unit: participants
Arm/Group | Enzastaurin-Cohort 2
Number analyzed (Participants) | 42
participants | 0

8. Secondary Outcome: Cohort 2 - PSA Velocity
Description: PSA velocity is defined as the rate of change in the PSA level during the first 2 and 3 months of the study.
Time Frame: baseline, 2 months and 3 months
Population: Participants in Cohort 2 with a valid baseline and at least one post-baseline PSA measurement within the first 2 and 3 months of treatment, respectively.
Measure: Mean (90% Confidence Interval); unit: nanograms per milliliter per year
Arm/Group | Enzastaurin-Cohort 2
Number analyzed (Participants) | 40
nanograms per milliliter per year
  PSA Velocity at 2 months | 0.30297 [0.13621 to 0.46972]
  PSA Velocity at 3 months | 0.26702 [0.10980 to 0.42423]

9. Secondary Outcome: Cohort 2 - Number of Participants With a Complete Response (CR) or Partial Response (PR) (Objective Response Rate)
Description: Objective responders in Cohort 2 met either CR or PR for composite criteria of PSA and RECIST. CR was defined as a decrease in PSA to an undetectable level (<0.2 ng/mL) confirmed by a second value at least 4 weeks apart and without clinical or radiographic evidence of disease per RECIST and normalization of bone scan. Bone only disease CR is normalization of bone scan with achievement of a nondetectable PSA confirmed 4-weeks after initial undetectable PSA. PR was defined as a decrease from baseline by 50% in PSA at any time during the study and confirmed by a second value at least 4 weeks apart and having at least a 30% decrease in sum of longest diameter of target lesions per RECIST and stable or improved bone scan.
Time Frame: baseline to first occurrence of tumor progression, skeletal event, symptomatic progression, or death (up to 31.3 months)
Population: Participants in Cohort 2 with a valid baseline and at least one post-baseline PSA assessment.
Measure: Number; unit: participants
Arm/Group | Enzastaurin-Cohort 2
Number analyzed (Participants) | 42
participants | 0

10. Secondary Outcome: Cohort 2 - Percentage of Participants With Progression Free Survival (PFS) at 6 Months and 12 Months
Description: Percentage of participants who did not meet the following criteria at 6 months and at 12 months: disease progression defined per RECIST for soft tissue lesions and/or the appearance of 2 or more new lesions on bone scan, or skeletal event (any pathological bone fracture, and/or need for palliative radiotherapy), or symptomatic progression (worsening ECOG performance status) and/or weight loss >10% from baseline and/or increase in analgesic consumption and pain, or death due to any cause. PFS was censored at the date of the most recent assessment for those who were still alive at the time of analysis and did not have evidence of tumor progression. Participants who took any subsequent systemic anticancer therapy prior to progression or death, PFS was censored at the date of the last objective progression-free disease assessment prior to the date of the subsequent systemic anticancer therapy. Percent=(number of participants meeting PFS criteria/number of randomized)x100.
Time Frame: 6 months and 12 months
Population: Participants in Cohort 2 who received at least 1 dose of enzastaurin. Two participants were censored.
Measure: Number; unit: percentage of participants
Arm/Group | Enzastaurin-Cohort 2
Number analyzed (Participants) | 42
percentage of participants
  6 month PFS rate | 3.0
  12 month PFS rate | 0.0

11. Secondary Outcome: Cohort 2 - Overall Survival
Description: Overall survival is the duration from enrollment to death. For participants who were alive, overall survival was censored at the last contact.
Time Frame: baseline to date of death from any cause (up to 69.6 weeks)
Population: Participants in Cohort 2 who received at least 1 dose of enzastaurin. Number of censored participants is 36.
Measure: Median (Full Range); unit: weeks
Arm/Group | Enzastaurin-Cohort 2
Number analyzed (Participants) | 42
weeks | NA [7.3 to 69.6] — Median was not defined due to high censoring rate (only 6 events).

12. Secondary Outcome: Cohort 2 - Duration of Response
Description: Duration of response was the date of first objective assessment of CR or PR to the date of first progression or death due to any cause. Progression of disease defined as:1) PSA progression: (a) in whom a 50% decline in PSA has not been achieved, defined as 25% increase over baseline or nadir whichever is lower and an increase in the absolute value of PSA level by 5 ng/mL and confirmed by another PSA at least 4 weeks apart, (b) in whom a 50% decline in PSA has been achieved, defined as 50% increase over the nadir and an increase in the absolute value of PSA level by 5 ng/mL and confirmed by another PSA level at least 4 weeks apart. 2) Objective Progression defined as radiographic evidence of metastatic disease irrespective of PSA value. 3) death due to any cause. Duration of response was censored on the date of discontinuation or last assessment for those participants who were alive without progression.
Time Frame: time of response to first occurrence of tumor progression, skeletal event, symptomatic progression, or death (up to 31.3 months)
Population: Zero participants were analyzed. Duration of response was not evaluable, as there were no participants with CR or PR in Cohort 2.
Arm/Group | Enzastaurin-Cohort 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Enzastaurin-Cohort 1 | Enzastaurin-Cohort 2
Serious Adverse Events (participants affected / at risk) | 2/31 | 12/42
Other Adverse Events (participants affected / at risk) | 29/31 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin-Cohort 1 (N=31) | Enzastaurin-Cohort 2 (N=42)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (2)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin-Cohort 1 (N=31) | Enzastaurin-Cohort 2 (N=42)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 13 (13)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 7 (7)
Fatigue (General disorders) | 12 (13) | 17 (18)
Oedema (General disorders) | 0 (0) | 6 (6)
Oedema peripheral (General disorders) | 4 (4) | 5 (6)
Pain (General disorders) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 3 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 3 (3)
Urine colour abnormal (Investigations) | 11 (11) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 12 (14)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypocholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (11)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (5) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hot flush (Vascular disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days